CLINICAL TRIAL: NCT04607122
Title: Interest of Low-dose Landiolol Administration After Cardiac Surgery for the Prevention of Postoperative Atrial Fibrillation
Brief Title: Prevention of Atrial Fibrillation by Low-dose Landiolol Administration After Cardiac Surgery
Acronym: LANDIPROTEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019/10; 2019-004829-25 (EudraCT Number)
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation; Cardiac Surgery
Keywords: Postoperative atrial fibrillation; Cardiac surgery; Landiolol hydrochloride; Low dose; Prophylactic administration
MeSH Terms: conditions — Atrial Fibrillation | interventions — landiolol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Landiolol group (Experimental): Landiolol infusion (2µg/kg/min) administrated after the surgery, on arrival at the ICU, until restoration of an effective oral beta-blocker treatment.
  Interventions: Drug: Landiolol
- Placebo group (Placebo Comparator): Saline solution infusion administrated after the surgery, on arrival at the ICU, until restoration of an effective oral beta-blocker treatment.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Landiolol — Continuous infusion of landiolol starting at 1 µg/kg/min and increasing every 10-15 minutes with incremental doses of 0.5 µg/kg/min up to 2 µg/kg/min by maintaining MAP ≥ 65 mmHg and HR ≥ 50/min.
  Other Names: Rapibloc
  Arms: Landiolol group
Drug: Saline — Continuous infusion of saline solution at the same rate as landiolol infusion.
  Other Names: Sodium chloride 0.9%
  Arms: Placebo group

SUMMARY:
Postoperative atrial fibrillation (POAF) is a common complication that occurs in 30-50% of patients after cardiac surgery and increases morbidity and mortality and hospital length of stay. During the perioperative period, the discontinuation of beta-blocker treatment is known to be a risk factor for developing POAF in patient undergoing cardiac surgery. Early beta-blocker reintroduction is associated with lower incidence of POAF. Unfortunately, side effects of currently available beta-blockers (including esmolol), such as low blood pressure and excessive bradycardia and/or their extended duration of action, limit their use in the post-operative period especially for prevention.

Landiolol, an ultra-short acting injectable beta-blocker, offers the advantage of significantly limiting low blood pressure events while increasing therapeutic efficacy in the treatment of POAF in cardiac and non-cardiac surgery. Landiolol, when used at low dose in the postoperative period, has been showed to reduce the incidence of POAF with no increased incidence of side effect as compared to standard of care. The limitation is that these promising data come from single center studies with limited samples and conducted exclusively in Japanese population. If landiolol is approved for use in the treatment of atrial fibrillation in non-Asian patients, there are no data on the prevention of POAF in cardiac surgery.

The objective of this multicenter, double-blind, randomized, placebo- controlled phase III trial is to confirm that landiolol postoperative infusion is associated with lower incidence of POAF without excess of adverse events as compared to standard of care in a non-Asian population after cardiac surgery with sternotomy.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group controlled, Landiolol vs Placebo (saline), phase III trial assessing the efficacy and the safety of landiolol postoperative treatment on POAF occurrence within 7 days of surgery in patients undergoing cardiac surgery with sternotomy.

Subjects are randomly assigned in a 1:1 ratio to receive either Landiolol or Placebo (saline). A stratification of the randomization is planned according to the hospital and the age of the patient (65 ≤ age ≤ 70 and age > 70).

A preventive treatment is infused during at least the first 24 hours after surgery (in ICU) to each patient included in the study until the optimal oral betablocker dose. Continuous infusion of landiolol at 2 µg/kg/min (1.2 ml/h, for a 60 kg patient) in Landiolol group or continuous infusion of saline (at 1.2 ml/h for a 60 kg patient) in Placebo group is administrated until restoration of an effective oral beta-blocker treatment.

Treatment:

Treatment is initiated after the surgery, on arrival at the ICU (Day-0) in the absence of a contraindication. The target of continuous intravenous infusion of landiolol is 2 µg/kg/min (1.2 ml/h for a 60 kg patient), or placebo (saline) at the same infusion rate as landiolol.

The modalities for initiating the treatment are as follows:

* No bolus is performed,
* Continuous infusion starting at the lowest dosage (1 µg/kg/min),
* Increasing in increments every 10 to 15 minutes until 2 µg/kg/min by maintaining a MAP ≥ 65 mmHg and HR ≥ 50/min.

Relay with oral betablocker treatment:

The relay with oral betablocker treatment, bisoprolol (1.25 mg x 2/day) for initial introduction (target HR < 100/min) or with the patient's preoperative beta-blocker in case of preoperative treatment, is resumed on Day-1 if possible or as soon as possible.

The dosage of landiolol can be reduced as follows:

* Within the first hour after the first dose of the alternative medicinal product has been administered, the infusion rate of landiolol should be reduced by one-half (e.g. from 2 to 1 µg/kg/min).
* After administration of the second dose of the alternative medicinal product (12 hours later), the patient's response should be supervised and if satisfactory control is maintained for a least one hour, the landiolol infusion can be discontinued.

Maximal duration of continuous intravenous treatment before oral betablocker relay is 5 days, exclusively administrated in ICU for safety reasons.

Precautions for patient safety:

The landiolol infusion should be decreased half and progressively re-increased every 15 min by step of 0.5 µg/kg/min and/or discontinued temporarily or permanently in case of:

* Bradycardia defined by HR < 50 /mim
* Hypotension defined by SAP < 90 mmHg or MAP < 65 mmHg
* Atrioventricular conduction treated by pacing
* Norepinephrine increase > 50% after introduction of landiolol infusion

In case of POAF event:

Patients will benefit from the usual care:

* Intravenous magnesium sulfate injection: 3 g over 1 hour
* Intravenous or per os treatment with amiodarone depending on patient's condition:

  * Intravenous: IV bolus of 300 mg over 1 hour; then IV infusion pump of 150-600 mg per day
  * Per os: loading dose with 4-6 tablets of 200 mg; then 2 tablets per day during one week
* If AF persists, cardioversion
* Anticoagulant therapy if required Treatment with landiolol or placebo is continued and the infusion rate is adjusted if needed as described above.

Primary endpoint: Continuous monitoring of heart rate is performed in ICU and POAF event > 5 minutes and/or requiring medical treatment and/or cardioversion is recorded during the ICU stay and reported.

ELIGIBILITY:
Inclusion Criteria:

* Non-Asian,
* Undergoing cardiac surgery with CPB,
* Left ventricular ejection fraction (LVEF) ≥ 40%,
* Having signed a written informed consent form,
* Affiliation to the social security system.

Preoperative Exclusion Criteria:

* Paroxystic or persistant atrial fibrillation before surgery,
* Preoperative contraindication to beta-blockers,
* Known hypersensitivity to landiolol,
* Severe conduction disorders (atrio-ventricular conduction block),
* A mental or linguistic inability to understand the study,
* Dying patient,
* Patient under protection of the adults (guardianship, curators or safeguard of justice),
* Patient included or planning to be included in another research protocol relating to medications.

Postoperative Exclusion Criteria:

- Postoperative contraindication to beta-blockers: severe sinus bradycardia requiring pacing, postcardiotomy low cardiac output requiring inotropic agents (noradrenaline being not considered as an inotropic agent), severe hypotension, severe acute pulmonary hypertension, reoperation for significant bleeding (> 200 ml/h), acute respiratory distress syndrome defined by increased oxygen dependence, a PaO2/FiO2 ratio < 200, polypnea > 30 /min, signs of respiratory distress (retractions, thoraco-abdominal asynchrony).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
POAF occurrence in Intensive Care Unit (ICU) | 7 days
  POAF event occurring from arrival to departure of the ICU assessed by continuous monitoring of heart rate (HR). POAF is defined as the occurrence of atrial fibrillation de novo, lasting more than 5 minutes (on the systematic reading of telemetry) and/or requiring specific medical treatment and/or cardioversion.

SECONDARY OUTCOMES:
Duration of POAF episode | 30 days
  Duration (in hours) of POAF episode categorized into five groups: POAF < 6h, POAF sustained ≥ 6h, POAF sustained ≥ 12h, POAF sustained ≥ 24h and POAF sustained ≥ 48h.
Day-30 POAF free days | 30 days
Need for cardioversion for POAF treatment | 30 days
Need for medical treatment for POAF treatment | 30 days
Delay between ICU admission and the first event of POAF | 30 days
Delay between the first event and the recidive of POAF | 30 days
Delay for discharge because of POAF event | 30 days
All-cause mortality | 30 days
In-ICU death | 30 days
In-hospital death | 30 days
Day-30 hospital free days | 30 days
  Length of hospital stay
Day-30 ICU free days | 30 days
  Length of ICU stay
Day-30 ventilator-free days | 30 days
Day-30 renal replacement therapy-free days | 30 days
Occurrence of major cardiovascular events | 30 days
  Cardiogenic shock, stroke or transient ischemic attack, seizure, cardiac arrest, myocardial infarction, Reoperation for bleeding, All-cause bleeding
Occurrence of drug adverse events | 7 days
  Bradycardia: HR < 50 bpm requiring heart pacing, Atrio-ventricular block requiring pacing, Severe hypotension: MAP < 50 mmHg requiring discontinuation of the protocol and specific treatment, Major ventricular arrhythmia requiring cardioversion.
Total hospital cost | 30 days
  Cost hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Julien Amour, MD, PhD, Principal Investigator — Hôpital Privé Jacques Cartier, Massy, France; Pierre Squara, MD, Study Chair — CMC Ambroise Paré, Neuilly-sur-Seine, France
Locations (3):
- France (3):
  - Hôpital Privé Jacques Cartier, Massy
  - CMC Ambroise Paré, Neuilly-sur-Seine
  - Centre Cardiologique du Nord, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amour J, Naudin C, Besnard A, Merzoug M, Laverdure F, Frossard B, Morichau-Beauchant T, Geri G, Squara P. Low dose of landiolol does not prevent postoperative atrial fibrillation after cardiac surgery in non-Asian patients: a multicentre randomised study. Br J Anaesth. 2026 Jan;136(1):65-73. doi: 10.1016/j.bja.2025.09.019. Epub 2025 Nov 6. PMID 41203473